CLINICAL TRIAL: NCT02523495
Title: The Clinical Outcome and the Exploration of Related Biomarkers of Target Therapy in Metastasis Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Chief physician, Huazhong University of Science and Technology
Other Study IDs: TJCC003-TTMCRC
Record Dates: First submitted 2015-08-04; First posted 2015-08-14 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms, Therapy-Associated
Keywords: Molecular Targeted Therapy; metastasis colorectal cancer; biomarker
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood

SUMMARY:
Through clinical observation and data statistics, conclude the clinical outcome of target therapy in metastasis colorectal cancer and explore some biomarkers that relate to target therapy.

DETAILED DESCRIPTION:
1. Establish a clinical database of patients who are diagnosed with metastasis colorectal cancer in tongji hospital.
2. Build a biological specimen banks of metastasis colorectal cancer through collecting blood samples from those patients who have reached an agreement with us.
3. Through clinical observation and data statistics, conclude the clinical outcome of target therapy in metastasis colorectal cancer.
4. To extract DNA from the blood and explore some biomarkers that related to target therapy in metastasis colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Metastasis colorectal cancer confirmed by histologically and radiography
2. Receive target therapy over half a year
3. Have a measurable lesions

Exclusion Criteria:

1. A history of other malignant tumors in five years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Metastasis colorectal cancer patients in Chinese Han population
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-06; Primary Completion 2020-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China